CLINICAL TRIAL: NCT05030480
Title: Prevalence of Chronic Kidney Disease and Associated Risk Factors Among Hypertensive Non-diabetic Patients in Ha'il Region, Saudi Arabia: A Cross-Sectional Study
Brief Title: Chronic Kidney Disease Among Hypertensive Patients in Ha'il, Saudi Arabia
Acronym: CKD
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Mohamed E Ghoniem, Associate Professor of Internal Medicine- Faculty of Medicine, Zagazig University
Other Study IDs: H-2020-206
Record Dates: First submitted 2021-08-20; First posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic kidney disease: eGFR values of less than 60 mL/min/1.73 m2
  Interventions: Diagnostic Test: renal functions
- Non-Chronic kidney disease: eGFR values more than 60 mL/min/1.73 m2
  Interventions: Diagnostic Test: renal functions

INTERVENTIONS:
Diagnostic Test: renal functions — urea, creatinine, GFR

SUMMARY:
Chronic kidney disease (CKD) is defined as persistent abnormalities of kidney structure or function for more than 3 months leading to a sustained reduction in glomerular filtration rate (GFR) and/or to the occurrence of kidney damage markers, such as albuminuria. [1] CKD is an emerging global public health problem, having significant morbidity and mortality costs on society. It is considered as an important component of the epidemic of non-communicable diseases in developed, as well as low-income/middle-income countries. [2] In the Kingdom of Saudi Arabia, CKD has been established as a major health issue in recent decades due to the growing incidence and prevalence of end stage kidney disease (ESKD) among the Saudi population. The overall prevalence of CKD was 5.7% in 2010. [3] In 2017, there were around two million cases of CKD and 3818 deaths due to CKD in Saudi Arabia in 2017. [4] A recent study also reported the overall prevalence of CKD stages 3 to 5 was 4.4% among the Saudi population. [5] The major consequences of CKD include disease progression and, subsequently, increased risk of cardiovascular disease.

DETAILED DESCRIPTION:
A cross-sectional study, enrolled 607 Saudi patients, of both sexes, registered for Ha'il University Medical Polyclinic, Ha'il city, Saudi Arabia, from October 6, 2020 to January 31, 2021. Patients eligible for inclusion in this study included those who were aged 18 years or older and were diagnosed with hypertension. Hypertension is defined as a systolic blood pressure (SBP) of 140 mm Hg or more, or a diastolic blood pressure (DBP) of 90 mm Hg or more, or taking antihypertensive medication or a positive self-reported history of hypertension (based on a response to the questions "have you ever been told you have high blood pressure" or "a past history of high blood pressure").[13] Exclusion criteria included pregnant or breastfeeding females; history of nephrotoxic drugs use and any case with known cause of CKD other than hypertension such as diabetes mellitus, polycystic kidney disease, obstructive uropathy or autoimmune diseases. Among 607 hypertensive patients who underwent health examinations, 175 patients met the exclusion criteria and were removed from the study. We also removed 40 patients from the remaining 432 individuals due to missing data, leaving 392 patients for analysis.Minimum sample required for this study was calculated using the formula: n = z2 [P (1 - P)/(D2)], confidence level at 95 % (z = 1.96), margin of error (D) is set at 0.05, and (P) is the prevalence of hypertension in adult Saudi population set as 25.5 %. (n = 292). Data was collected through an interview questionnaire. The questionnaire included sociodemographic variables (age, sex, height, weight, BMI and smoking habit), hypertension (duration and drugs taken), as well as other chronic comorbidities in addition to previous family history of renal diseases. This is in addition to the laboratory investigations and radiological reports collected from the participants during the interview.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for inclusion in this study included those who were aged 18 years or older and were diagnosed with hypertension

Exclusion Criteria:

* pregnant or breastfeeding females; history of nephrotoxic drugs use and any case with known cause of CKD other than hypertension such as diabetes mellitus, polycystic kidney disease, obstructive uropathy or autoimmune diseases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A cross-sectional study, enrolled 607 Saudi patients, of both sexes, registered for Ha'il University Medical Polyclinic, Ha'il city, Saudi Arabia, from October 6, 2020 to January 31, 2021. Patients eligible for inclusion in this study included those who were aged 18 years or older and were diagnosed with hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 392 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
PREVALANCE AND REISK FACTORS | 3 MONTHS
  Prevalence of Chronic Kidney Disease and Associated Risk Factors among hypertensive non-diabetic patients

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ha'il, Ha'il, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided